CLINICAL TRIAL: NCT02269787
Title: TeleMonitoring to Improve Substance Use Disorder Treatment After Detoxification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRE 12-010
Record Dates: First submitted 2014-10-03; First posted 2014-10-21 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Enhanced Telephone Monitoring; Usual Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Telephone Monitoring (Experimental): Detox inpatients in the ETM condition will be expected to complete one 15-minute telephone call per week for 12 weeks.
  Interventions: Behavioral: Enhanced Telephone Monitoring
- Usual Care (No Intervention): Patients in the usual care condition will receive the care they would receive in the absence of a research project.

INTERVENTIONS:
Behavioral: Enhanced Telephone Monitoring — Detox inpatients in the ETM condition will be expected to complete one session while in detox and one 15-minute telephone call per week for 12 weeks (plus usual care).
  Other Names: ETM
  Arms: Enhanced Telephone Monitoring

SUMMARY:
This research program is intended to improve the treatment engagement and outcomes of Veterans who receive inpatient detoxification, and decrease their use of VA inpatient and emergency department services. It is intended to increase the use of substance use disorder care and 12-step mutual-help groups to benefit recovery, reduce rehospitalizations, and reduce costs for VA.

DETAILED DESCRIPTION:
Annually, about 25,000 Veterans receive inpatient detoxification (detox) for substance use disorders (SUDs). Detox is not SUD treatment; it is the medical management of withdrawal to prevent complications, which may be fatal. Detox inpatients who enter SUD treatment and peer-based mutual-help groups (e.g., Alcoholics Anonymous) have much better outcomes (less substance use, HIV/HCV risk behaviors, homelessness, rehospitalizations, Emergency Department visits) than those who do not. However, because of their unique characteristics (severe and chronic addictions, co-morbidities, lack of resources, self- and provider-perceptions as unsuitable for treatment), most Veterans discharged from inpatient detox do not enter SUD treatment. For many Veterans, a pattern of repeated inpatient detox, with each episode incurring a higher risk of overdose, occurs. Therefore, in its Uniform Services Handbook, Mental Health Operations places major emphasis on increasing the rate of SUD treatment initiation and engagement following detox to benefit Veterans' outcomes and prevent more use of costly health care.

The primary objective of this project is to implement and evaluate Enhanced Telephone Monitoring (ETM) as a new and innovative telehealth intervention to facilitate the transition from inpatient detox to SUD specialty treatment (residential, outpatient, pharmacotherapy), thereby improving Veterans' outcomes and decreasing VA health care costs. In a randomized trial at two sites (VA Palo Alto and Boston), investigators hypothesize that patients receiving ETM, compared to patients in usual care (UC), will be more likely to enter and engage in SUD treatment and mutual-help, have better SUD and related outcomes, and have fewer and delayed acute care episodes. This project will also conduct a formative evaluation of how to implement ETM VA-wide, focusing on diverse subgroups of Veterans. Further, it will conduct a Budget Impact Analysis (BIA) to determine the impact of ETM on total costs of VA care. Investigators hypothesize that the higher costs associated with ETM (because patients will engage in SUD treatment) will be more than offset by its lower costs of acute care.

Patients in the ETM condition will receive an in-person session while in detox, followed by coaching over the telephone for 3 months after discharge. The intervention will incorporate Motivational Interviewing, and Contracting, Prompting, and Reinforcing, to provide support while waiting for treatment, and facilitate entry into treatment and mutual-help, and improved responses to crises. Patients will be assessed at baseline and 3 and 6 months post-discharge for outcomes and non-VA health care; VA health care will be assessed with VA databases. GLMM analyses will be conducted to compare the UC and ETM groups on course of outcomes over time. The formative evaluation to inform the implementation of ETM will use the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework. Semi-structured interviews will be conducted with inpatient detox staff and patients to yield facilitators of ETM implementation and modifiable barriers with associated action plans. For the BIA, costs of ETM will be measured through microcosting methods. For patients in both the ETM and UC groups, all inpatient, residential, outpatient, and pharmacy care will be measured from VA utilization and cost files.

In summary, Mental Health Operations is committed to eradicating the dangerous, costly pattern of Veterans obtaining inpatient detox services but not receiving the SUD treatment they need. Telehealth interventions, a promising way to improve treatment access and outcomes by SUD patients, have not been utilized with the challenging population of detox inpatients before. In accordance with others in this CREATE, this project will help to accomplish Mental Health Operations' goal of implementing the Uniform Handbook by increasing Veterans' access to, engagement in, and benefit from, SUD treatment services, particularly among Veterans who are using VA medical services and need SUD services but are not receiving them.

ELIGIBILITY:
Inclusion Criteria:

* Beginning an episode of inpatient detoxification at the Boston or Palo Alto Veterans Affairs medical facilities, and
* have ongoing access to cell phone or land line telephone

Exclusion Criteria:

* Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Timko, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Telephone Monitoring: Detox inpatients in the ETM condition will be expected to complete one 50-minute individual session while in detox and one 15-minute telephone call per week for 12 weeks (plus usual care).
- Usual Care: Detox inpatients in the usual care condition will receive the care they would receive in the absence of a research project.
Period: Overall Study
Arm/Group | Enhanced Telephone Monitoring | Usual Care
Started | 148 | 150
Completed | 126 | 140
Not Completed | 22 | 10
Not completed — Lost to Follow-up | 20 | 6
Not completed — Death | 2 | 3
Not completed — Incapacitated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Telephone Monitoring | Usual Care | Total
Number analyzed (Participants) | 148 | 150 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.9) | 48.9 (13.5) | 50.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 141 | 142 | 283
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 112 | 113 | 225
  Other | 36 | 37 | 73
Married [Count of Participants; unit: Participants] | 28 | 26 | 54
Years education [Mean (Standard Deviation); unit: years] | 13.0 (1.8) | 13.3 (1.9) | 13.1 (1.8)
Employed [Count of Participants; unit: Participants] | 46 | 55 | 101
Homeless [Count of Participants; unit: Participants] | 23 | 20 | 43
Detoxification, lifetime [Count of Participants; unit: Participants] | 145 | 145 | 290
Attended 12-step meeting (past 3 months) [Count of Participants; unit: Participants] | 81 | 79 | 160
Number of meetings (past 3 months) [Mean (Standard Deviation); unit: meetings] | 7.0 (14.3) | 8.6 (15.8) | 8.5 (22.7)
Treatment, lifetime [Count of Participants; unit: Participants] | 91 | 88 | 179
Treatment, 30 days [Count of Participants; unit: Participants] | 16 | 14 | 30
ASI, Alcohol severity [Mean (Standard Deviation); unit: units on a scale] — ASI composite scores were produced from sets of items that were standardized and summed to provide internally consistent evaluations of patient status in the problem areas (McLellan et al., 2006). They range from 0 to 1, with higher scores indicating poorer outcomes. Alcohol Severity is a composite score for the ASI alcohol dimension which measures the severity of the problem in that area over the past 30 days.
  units on a scale | .564 (.290) | .565 (.290) | .565 (.299)
ASI, Drugs severity [Mean (Standard Deviation); unit: units on a scale] — ASI composite scores were produced from sets of items that were standardized and summed to provide internally consistent evaluations of patient status in the problem areas (McLellan et al., 2006). They range from 0 to 1, with higher scores indicating poorer outcomes. Drug Severity is a composite score for the ASI drug dimension which measures the severity of the problem in that area over the past 30 days.
  units on a scale | .134 (.151) | .125 (.157) | .130 (.154)
ASI, Psychiatric [Mean (Standard Deviation); unit: units on a scale] — ASI composite scores were produced from sets of items that were standardized and summed to provide internally consistent evaluations of patient status in the problem areas (McLellan et al., 2006). They range from 0 to 1, with higher scores indicating poorer outcomes. Psychiatric is a composite score for the ASI psychiatric dimension which measures the severity of the problem in that area over the past 30 days.
  units on a scale | .479 (.226) | .490 (.236) | .485 (.231)
Days used alcohol (past 30 days) [Mean (Standard Deviation); unit: days] | 16.0 (10.7) | 15.3 (10.8) | 15.7 (10.8)
Days used opioids (past 30 days) [Mean (Standard Deviation); unit: days] | 5.1 (11.0) | 5.6 (11.7) | 5.3 (11.3)
Serious ideas suicide (past 30 days) [Count of Participants; unit: Participants] | 47 | 49 | 96
Attempted suicide (past 30 days) [Count of Participants; unit: Participants] | 15 | 15 | 30
BAM, Alcohol and drug use [Mean (Standard Deviation); unit: units on a scale] — Brief Addiction Monitor (which is required in VA for measurement based substance use disorder care) yields two composite scores referring to the past 30 days. Alcohol and drug use is the sum of three items, i.e., number of days drank alcohol; had at least 5 drinks (if a man) or at least 4 drinks (if a woman); and used any illegal/street drugs or abused any prescription medications (for each, 0=0 days, to 4=16-30 days, i.e. higher the mean, more days used substances).
  units on a scale | 7.2 (3.1) | 7.0 (2.9) | 7.1 (3.0)
BAM, Risk factors [Mean (Standard Deviation); unit: units on a scale] — Brief Addiction Monitor (which is required in VA for measurement based substance use disorder care) yields two composite scores referring to the past 30 days. Risk factors is the sum of five items, e.g., physical health (0=excellent, 4=poor); number of nights having trouble falling or staying asleep (0=0, 4=16-30 days); in any situations or with any people that might increase risk for using alcohol or drugs (0=0, 4=16-30 days, higher the mean, worse the outcome/higher risk for substance use).
  units on a scale | 15.0 (4.6) | 15.6 (4.3) | 15.3 (4.5)
Self-efficacy, Confidence [Mean (Standard Deviation); unit: units on a scale] — Self-efficacy was assessed with the Brief Situational Confidence Questionnaire (Breslin, Sobell, Sobell, & Agrawal, 2000). Eight items asked patients to rate their level of confidence (0% 'not at all confident' to 100% 'totally confident') in resisting drinking and using drugs as a response to different types of situations (e.g., unpleasant emotions, social pressure to drink/use), and then responses were averaged such that higher scores indicate more self-efficacy (Cronbach's alpha = .91, .92, and .91 at baseline and 3 and 6 months, respectively).
  units on a scale | 62.1 (29.0) | 58.4 (26.7) | 60.2 (27.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Had an Additional Inpatient Detoxification
Description: Percent that had (yes) an additional inpatient detoxification 6 months following baseline assessment- additional inpatient detoxification was dichotomous, yes or no.
Time Frame: 6-month follow-up
Population: Of 298 baseline participants, 266 participated in follow-up at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Telephone Monitoring | Usual Care
Number analyzed (Participants) | 126 | 140
Participants | 33 | 47

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Enhanced Telephone Monitoring | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/148 | 3/150
Serious Adverse Events (participants affected / at risk) | 0/148 | 1/150
Other Adverse Events (participants affected / at risk) | 0/148 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Telephone Monitoring (N=148) | Usual Care (N=150)
Incapacitation (General disorders) | 0 (0) | 1 (1) — Too incapacitated by poor health to complete follow-up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT02269787/Prot_SAP_000.pdf